CLINICAL TRIAL: NCT02341300
Title: Use of Cast Iron Pots to Improve Maternal Anemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original investigator has left the institution.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1310014372
Record Dates: First submitted 2014-07-30; First posted 2015-01-19 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Iron-deficiency Anemia
Keywords: Pregnancy; Cast-Iron pots; Iron-deficiency anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast-Iron Pot (Experimental): The treatment arm will receive a 12 inch pre seasoned cast iron pot
  Interventions: Device: Cast Iron Pot
- Aluminum Pot (Placebo Comparator): 12 inch nonstick aluminum fry pan
  Interventions: Device: Alumnium Pot

INTERVENTIONS:
Device: Cast Iron Pot — Cast iron pot
  Other Names: Lodge L10SK3 12" Pre-Seasoned Cast Iron Skillet
  Arms: Cast-Iron Pot
Device: Alumnium Pot — Aluminum Skillet
  Other Names: Alumnium Skillet
  Arms: Aluminum Pot

SUMMARY:
Anemia of pregnancy is defined as a hemoglobin concentration of less than 11 g/dL in the first and third trimesters, and less than 10.5 g/dL in the second trimester. The rates of anemia are variable and depend largely on preexisting iron stores and supplementation. Estimates from the World Health Organization report that 35% to 75% of pregnant women in developing countries and 18% of women from industrialized countries are anemic. Maternal anemia is associated with an increased risk of preterm birth, low birthweight, and small for gestational age infants. Many studies have shown improvement in these outcomes with maternal iron supplementation in cases of iron-deficiency anemia. Mounting evidence also indicates that maternal iron deficiency in pregnancy reduces fetal iron stores, perhaps well into the first year of life.

Anemia in pregnancy can also impact maternal morbidity and mortality. Viteri reported that anemic pregnant women are at greater risk of death during the perinatal period and that anemia is the major contributory or sole cause of death in 20-40% of the 500,000 maternal deaths per year.

The need for iron averages close to 1000mg in a typical singleton gestation. This amount considerably exceeds the iron stores of most women and will result in iron-deficiency anemia unless supplemental iron is taken. One problem with iron supplement use is compliance, secondary to adverse effects such as constipation and nausea. Research on the use of cast iron pots in decreasing the incidence of iron-deficiency anemia in non-pregnant women has been promising. These studies have demonstrated good compliance with no reported adverse effects. The aim of our study is to determine if providing anemic women in the first trimester of pregnancy with a cast iron pot will decrease the incidence of anemia later in pregnancy.

Hypothesis: Cooking in cast iron pots will increase hematocrit levels in pregnancy.

DETAILED DESCRIPTION:
Research Question: Will the addition of cast iron pots to the standard of care (nutrition counseling, food recall, prenatal vitamin, +/- iron and vit c) improve the hematocrit of pregnant women with anemia? Study Intervention: To provide a cast iron pot to those pregnant women with anemia who are randomized to intervention group and an aluminum pot to those women in the control group. Women will be blinded to their allocation. Women with a qualifying hemoglobin will meet with our nutritionist (as they would if not enrolled in the study), and she will perform a standardized 24 hour food recall and nutrition counseling according to the standard of care, as well as perform written informed consent. The 24 hour food recall will be submitted to the manufacturer (Nutrition Quest) to calculate the baseline iron intake of each subject. Subjects will be enrolled only if they can agree to incorporate the provided pot into their cooking (in any capacity) 3x/week. Subjects will be called 1x/month and asked about the frequency of pot use over the past month as well as their compliance with iron and vitamin C supplements, if prescribed. Subjects will then also be contacted postpartum to determine satisfaction with the intervention.

Outcome measure: We will be looking at hemoglobin levels in the first, second, and third trimester as well as postpartum (which are all routinely collected labs in pregnancy). Ferritin will be added along with routine labs at approximately 19 weeks as this is often performed in the workup of anemia. No labs outside of routine maternal labs will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of any age in their first trimester of pregnancy with anemia defined as a Hemoglobin less than 11 and/or a hematocrit less than 33
* Willingness and ability to cook in provided cast iron pot at least 3x/week
* Singleton gestations

Exclusion Criteria:

* Any secondary cause of anemia including inherited and acquired hemolytic anemias (sickle cell disease, thalessemia, malaria, etc) Inability or unwillingness to try to use cast iron pot approximately 3x/week
* Women with severe chronic illness and high likelihood of preterm birth and/or expected long-term hospitalizations during pregnancy. Multifetal gestations

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Increased hematocrit in second and third trimesters of pregnancy | 28 weeks (2nd and 3rd trimesters of pregnancy)

SECONDARY OUTCOMES:
Compliance assessment | postpartum, after ~30 weeks
  We will assess compliance with iron/aluminium pot use at the conclusion of the study
Incidence of adverse effects | Monthly phone surveys for 28 weeks
  Will contact patients to assess incidence of adverse effects of iron including constipation
Satisfaction | Monthly phone surveys for 28 weeks
  Will contact patient monthly to assess satisfaction with study intervention
Maternal anemia postpartum | postpartum, after ~30 weeks
  Will assess subjects need for transfusion and/or symptoms of anemia (dizziness, lightheadedness) postpartum
Neonatal outcomes | postpartum, at ~30 weeks
  Will follow up neonatal outcomes to assess for prematurity and/or low birthweight

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chasen, MD, Principal Investigator — New York Presbyterian Hospital Weill Cornell
Locations (1):
- New York Prebyterian Hospital Weill Cornell, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data may be shared. No biologic specimens are being collected in this study